CLINICAL TRIAL: NCT06226597
Title: Fitbit Device Use in Overweight Pregnant Women to Improve Adherence to Gestational Weight Gain Guidelines
Brief Title: Fitbit Device Use in Overweight Pregnancy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Laura Mroue, Principal Investigator, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1101840
Record Dates: First submitted 2024-01-03; First posted 2024-01-26 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Pregnancy Weight Gain; Overweight and Obesity
Keywords: Pregnancy; Overweight or obese; Physical activity; Sleep in Pregnancy
MeSH Terms: conditions — Gestational Weight Gain; Overweight; Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fitbit monitoring (Experimental): Individuals in this arm will wear a fitbit device consistently throughout the duration of their pregnancy, and monitor fitbit data using a platform that connects to their phone. The remainder of prenatal care will be per standard procedure.
  Interventions: Device: Fitbit device
- Routine prenatal care (No Intervention): Individuals in this arm will receive standard prenatal care without the addition of wearing a fitbit device.

INTERVENTIONS:
Device: Fitbit device — Daily use of a fitbit wearable activity tracker device.
  Arms: Fitbit monitoring

SUMMARY:
There are set guidelines for weight gain developed by the Institute of Medicine in pregnancy but about three quarters of women gain an inappropriate weight during pregnancy. Many studies have assessed ways to decrease weight gain in these women who gain excess weight, usually through a combination of diet and exercise. Still, often these interventions are difficult to implement, expensive, or have low acceptability. Wearable Fitbit devices have been on the market for years and slowly becoming more inexpensive and easier to use.

Previous studies on non-pregnant women have shown that using the device can help reduce weight gain. In addition, small studies in pregnant women have shown they are accurate for measuring steps and have high acceptability and retention rates. The ability of the Fitbit to assess metrics of sleep including sleep duration and quality will also be assessed.

This project aims to provide overweight and obese pregnant women at the beginning of their pregnancy with the Fitbit device and with regular follow-up to assess if there is effectiveness in increasing the rate of women who meet weight gain guidelines compared to women without the device along with measuring aspects of sleep.

DETAILED DESCRIPTION:
This is a prospective randomized control trial study. This study aims to assess the relationship between physical activity and sleep metrics in pregnant women as measured using the Fitbit device and the ability to meet Institute of Medicine weight gain guidelines during pregnancy. The hypothesis of the study is that self-realization and monitoring of activity using the Fitbit will encourage the wearer to be increasingly physically active and assist in meeting weight gain guidelines. This study is performed in conjunction with the University of Arizona sensor lab utilizing the MyDataHelps platform which will assist with collection of data from each participant's Fitbit device and subsequent analysis. Mydatahelps is an easily customizable data collection platform that helps researchers collect participant data in a secure HIPAA compliant manner. They are an external company but have no input in the construction of the project This study will have two arms: one with Fitbit wearers and a control arm for routine prenatal care. Compared to control participants who will not have a Fitbit device, we hypothesize that utilization of the Fitbit device will be effective in helping overweight and obese pregnant women meet Institute of Medicine weight gain guidelines.

The primary endpoint is gestational weight gain throughout pregnancy. Weight will be measured pre-pregnancy, at recruitment, 28 weeks, delivery, and 6 weeks postpartum.

Secondary endpoints will also be measured and include:

1. Acceptability of device and loss to follow-up
2. Obstetrical outcomes include rate of developing gestational diabetes, gestational hypertension and preeclampsia, preterm delivery, cesarean delivery rate, intrauterine growth restriction, and macrosomia
3. Neonatal outcomes, including birth weight and admission to NICU
4. Fitbit outcome data, including steps taken, calories burned, sleep duration and Fitbit derived sleep quality
5. Questionnaire data: Global Physical Activity Questionnaire (GPAQ), Cambridge Worry Scale and Pittsburgh Sleep Quality Index at baseline, 28 weeks and delivery

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Currently pregnant with a singleton pregnancy
* Pre-pregnancy body mass index over 25
* Owns and uses a smartphone
* Agreeable to participate in the study by wearing a fitbit device consistently (day and night) for the duration of pregnancy

Exclusion Criteria:

* Multiple gestations
* Beyond the first trimester at time of initial enrollment
* Known maternal cardiac disease
* Pre-gestational diabetes
* High risk of preterm labor
* Any contraindications to exercise
* Unwilling to wear device consistently or share tracked data

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-02-08 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Gestational weight gain during pregnancy | From pre-pregnancy or initial prenatal visit until 6 weeks postpartum
  Weight will be measured pre-pregnancy, at recruitment (ideally initial prenatal visit), 28 weeks gestation, at delivery and 6 weeks postpartum

SECONDARY OUTCOMES:
Number of patients reporting adverse events related to device | Through duration of participation, average of 8-9 months
  Tolerability of wearing the device consistently, any adverse effects
Number of patients lost to follow-up | 18 months
  Individuals that discontinue follow-up or study inclusion
Incidence of intrauterine growth restriction | At delivery
  Number of pregnancies affected by intrauterine growth restriction
Incidence of fetal macrosomia | At delivery
  Number of pregnancies affected by fetal macrosomia
Incidence of gestational hypertension | At delivery
  Number of patients who develop gestational hypertension in pregnancy
Incidence of gestational diabetes | At delivery
  Number of patients who develop gestational diabetes in pregnancy
Incidence of preeclampsia | At delivery
  Number of patients who develop preeclampsia in pregnancy
Incidence of preterm delivery | At delivery
  Number of patients who experience preterm delivery
Incidence of cesarean delivery | At delivery
  Number of patients who have cesarean delivery
Neonatal birth weight | At delivery
  Neonatal birth weight in grams
Incidence of NICU admission | At delivery
  Number of fetuses requiring admission to neonatal ICU care
Average number of daily steps taken per individual | At delivery
  Average number of daily steps taken per individual as recorded by fitbit device
Calories burned per individual | At delivery
  Daily calories burned per individual, as measured by fitbit device, in kcal
Daily sleep duration | At delivery
  Daily and average sleep duration in hours per individual, as measured by fitbit device
Fitbit derived sleep quality | At delivery
  Fitbit device determined nightly sleep score
Global Physical Activity Questionnaire (GPAQ) score | At initial enrollment, 28 weeks gestation and delivery
  Questionnaire data
Cambridge Worry Scale score | At initial enrollment, 28 weeks gestation and delivery
  Questionnaire data
Pittsburg Sleep Quality Index score | At initial enrollment, 28 weeks gestation and delivery
  Questionnaire data

CONTACTS AND LOCATIONS:
Overall Officials: Laura Mroue, MD, Principal Investigator — University of Arizona
Locations (1):
- Banner University Medical Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon request and approval by the study team, IPD may be shared with other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within 6 months of study publication.
Access Criteria: Access will be available by contacting the study PI for approval.

REFERENCES:
- [Background] Deputy NP, Dub B, Sharma AJ. Prevalence and Trends in Prepregnancy Normal Weight - 48 States, New York City, and District of Columbia, 2011-2015. MMWR Morb Mortal Wkly Rep. 2018 Jan 5;66(51-52):1402-1407. doi: 10.15585/mmwr.mm665152a3. PMID 29300720
- [Background] Rasmussen KM, Catalano PM, Yaktine AL. New guidelines for weight gain during pregnancy: what obstetrician/gynecologists should know. Curr Opin Obstet Gynecol. 2009 Dec;21(6):521-6. doi: 10.1097/GCO.0b013e328332d24e. PMID 19809317
- [Background] Goldstein RF, Abell SK, Ranasinha S, Misso M, Boyle JA, Black MH, Li N, Hu G, Corrado F, Rode L, Kim YJ, Haugen M, Song WO, Kim MH, Bogaerts A, Devlieger R, Chung JH, Teede HJ. Association of Gestational Weight Gain With Maternal and Infant Outcomes: A Systematic Review and Meta-analysis. JAMA. 2017 Jun 6;317(21):2207-2225. doi: 10.1001/jama.2017.3635. PMID 28586887